CLINICAL TRIAL: NCT03461666
Title: A Randomized, Open Label, Sleep Hygiene Controlled 6-Week Study to Compare the Efficacy of Four (CBT-I, FOA, Combined CBT-I and FOA and Sleep Hygiene) Different Behavioral Approaches for the Treatment of Adult Subjects With Insomnia
Brief Title: Comparison of Efficacy of Behavioral Approaches for Treatment of Insomnia
Acronym: CEBATI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention. COVID Complications.
Sponsor: Pacific Institute of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PSPC-17-01
Record Dates: First submitted 2017-12-22; First posted 2018-03-12 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Primary Insomnia
Keywords: Primary insomnia; Behavioral treatment of primary insomnia; Focus of attention; cognitive behavioral therapy for insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Behavior Therapy-Insomnia (Active Comparator): Participants receive 6 one hour in person behavioral psycho-intervention sessions from a treatment provider.
  Interventions: Behavioral: Cognitive Behavior Therapy-Insomnia; Behavioral: Focus of Attention; Behavioral: Combined-CBT-I and FOA Group; Behavioral: Sleep Hygiene
- Focus Of Attention (Active Comparator): Participants receive 6 one hour in person behavioral psycho-intervention sessions from a treatment provider.
  Interventions: Behavioral: Cognitive Behavior Therapy-Insomnia; Behavioral: Focus of Attention; Behavioral: Combined-CBT-I and FOA Group; Behavioral: Sleep Hygiene
- Combined-CBT-I and FOA Group (Active Comparator): Participants receive 6 one hour in person behavioral psycho-intervention sessions from a treatment provider.
  Interventions: Behavioral: Cognitive Behavior Therapy-Insomnia; Behavioral: Focus of Attention; Behavioral: Combined-CBT-I and FOA Group; Behavioral: Sleep Hygiene
- Sleep Hygiene (Active Comparator): Participants receive 6 one hour in person behavioral psycho-intervention sessions from a treatment provider.
  Interventions: Behavioral: Cognitive Behavior Therapy-Insomnia; Behavioral: Focus of Attention; Behavioral: Combined-CBT-I and FOA Group; Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy-Insomnia — Behavioral Psycho-intervention education therapy.Face to Face, Six sessions, one hour each.
Behavioral: Focus of Attention — Behavioral Psycho-intervention education therapy.Face to Face, Six sessions, one hour each.
Behavioral: Combined-CBT-I and FOA Group — Behavioral Psycho-intervention education therapy.Face to Face, Six sessions, one hour each.
Behavioral: Sleep Hygiene — Behavioral Psycho-intervention education therapy.Face to Face, Six sessions, one hour each.

SUMMARY:
This study compares the efficacy of four different types (Cognitive Behavior Therapy for Insomnia (CBT-I); Focus of Attention (FOA); Combined CBT-I and FOA; and Sleep Hygiene (control group) for the treatment of insomnia. This study is a randomized, open label study, and the participants are asked to assess the benefits they get from the intervention. This study involve 6 weekly in person one-to-one sessions after screening and completion of the 1-week, 3-month, 6-month and 12-month follow-up assessment. The trained study staff will administering the treatment. The Research Department will administer the outcome measures. The review of insomnia improvement will be assessed at at end of treatment, 3 months, 6 months and 12 months follow-up.

DETAILED DESCRIPTION:
This study compares the efficacy of four different types (Cognitive Behavior Therapy for Insomnia (CBT-I), Focus of Attention (FOA), Combined CBT-I and FOA and Sleep Hygiene) of therapies approaches for the treatment of insomnia. This study is a randomized, open label study, the participants are asked to review the benefits they get from the intervention. This study involve 6 weekly sessions after screening and completion of the end of treatment, 3-month, 6-month and 12-month follow-up assessment. The trained study staff will administer study scales during therapy session. The subjective review of insomnia improvement will be assessed at end of treatment, 3 months, 6 months and 12 months follow-up assessment. Subjects are adult who meet, DSM-5 the diagnostic criteria for primary Insomnia.

Inclusion/Exclusion criteria to be assessed at Screening (Visit 1) and Visit 2. For those found eligible who complete the study, participation will include Screening (Visit 1), 6 weekly sessions after screening, and completion of the post-treatment and 6-month followup assessment.

Once subject sign the consent form, subject will be asked inclusion and exclusion criteria and will be given details about the study as per protocol.

Those eligible will be randomly assigned to one of four behavioral treatment approaches. The participant will have six weekly one hour in person sessions in which the assigned treatment will be administered. The participant will be assessed at the end of treatment and again at 6 month followup.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients who are 18 or older to 72 years. Insomnia Severity Index > or = 10
* Meet diagnostic criteria for Insomnia Disorder per DSM-5 Willing and able to sign Informed consent form Not planning on moving away from the area for the subsequent 12 weeks.

Exclusion Criteria:

* Participants who answer "yes" to any of the following will be excluded:
* Females who are lactating or who are pregnant
* Night shift workers, and individuals who nap 3 or more times per week over the preceding month
* Consumption of caffeine beverages (i.e. tea, coffee, or cola) comprising usually more than 5 cups or glasses per day
* Participation in another trial for insomnia
* Persons unable to complete the study questionnaires and psychological tests
* Persons who are unable to participate for the entire duration of the study, or in the opinion of the investigators, are likely to be non-compliant with the obligations inherent in the trial participation
* Persons self-describing with severe anxiety or severe depression (BDI score of 29 or higher) or severe anxiety (BAI score of 36 or higher).
* Persons with a history of epilepsy, seizures, or dementia
* Any significant, severe or unstable, acute or chronically progressive medical or surgical condition
* Serious head injury or stroke within the past year
* Current alcohol or substance abuse/dependence (must have >90 days of sobriety)
* Presence of other neurological disorders (e.g., multiple sclerosis, Parkinson's Disease)
* Presence of an untreated or unstable medical or psychiatric comorbid condition (e.g., major depressive disorder or psychotic disorder requiring admission within the last two years). People using psychotropic medication, hypnotic or sedative medications may be included if they are on a stable dosage for the last 2 months prior to the study, if the dose remains stable throughout the study, and if the medication is judged to not interfere with the study outcomes.
* Currently on medications known to produce insomnia (e.g., stimulants)
* Sleep apnea (AHI >15) or previous diagnosis of sleep apnea. Study participants who use a continuous positive airway pressure (CPAP) device for sleep apnea will be eligible for participation if they are below the apnea/hypopnea cutoff while using CPAP and agree to use the device during study participation.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Self Report Sleep Measures | through study completion, an average of 1 year
  SRSM: assess overall quantity of sleep satisfaction on the Self Report Sleep Measures.

SECONDARY OUTCOMES:
Insomnia Severity Index | through study completion, an average of 1 year
  ISI: assess the severity of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Max Hines, Ph.D, Principal Investigator — Puget Sound Psychiatry center
Locations (2):
- United States (2):
  - Puget Sound Psychiatric Center, Bothell, Washington
  - Puget Sound Psychiatry Center, Bothell, Washington

IPD SHARING:
Plan to Share IPD: No
Finding to present in peer review journals

REFERENCES:
- [Result] Becher AK, Hohne M, Axmacher N, Chaieb L, Elger CE, Fell J. Intracranial electroencephalography power and phase synchronization changes during monaural and binaural beat stimulation. Eur J Neurosci. 2015 Jan;41(2):254-63. doi: 10.1111/ejn.12760. Epub 2014 Oct 25. PMID 25345689
- [Result] Cahn BR, Polich J. Meditation states and traits: EEG, ERP, and neuroimaging studies. Psychol Bull. 2006 Mar;132(2):180-211. doi: 10.1037/0033-2909.132.2.180. PMID 16536641

DOCUMENTS (2):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03461666/Prot_002.pdf
  • Informed Consent Form (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03461666/ICF_004.pdf